CLINICAL TRIAL: NCT00006099
Title: Pilot Trial of Humanized 3S193 Monoclonal Antibody (hu3S193) in Presurgical Patients With Ovarian Cancer
Brief Title: Monoclonal Antibody Therapy in Treating Patients Scheduled for Surgery to Remove Ovarian Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low study accrual
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000068107; MSKCC-00047 (Other: Memorial Sloan-Kettering Cancer Center); NCI-G00-1828 (Other: National Cancer Institute); LUD1998-013 (Other: Ludwig Institute for Cancer Research)
Record Dates: First submitted 2000-08-03; First posted 2003-12-23 (Estimated); Results first posted 2021-08-12 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Ovarian Cancer
Keywords: ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Hu3S193 monoclonal antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intraperitoneal (IP) Infusion of 111In-hu3S193 (Experimental): Hu3S193 was administered intraperitoneally at a dose of 5 mg radiolabeled with 5 millicurie (mCi) of 111In.
  Patients received 10 mCi 99mTc-sulphur colloid IP administered in 500 ml of normal saline to assure the absence of any loculation or heterogeneous distribution of radioactivity in the peritoneal cavity. A paracentesis catheter was inserted and the hu3S193 was diluted in 100 mL of 5% human serum albumin and administered as a continuous intraperitoneal infusion over 30 minutes. This was followed immediately by 900 mL of normal saline.
  Interventions: Biological: Monoclonal antibody hu3S193
- Intravenous Infusion of 111In-hu3S193 (Experimental): Hu3S193 was to be administered intravenously at a dose of 5 mg radiolabeled with 5 millicurie (mCi) of 111In, diluted in 100 mL of 5% human serum albumin and administered over a 30 minute period.
  Interventions: Biological: Monoclonal antibody hu3S193

INTERVENTIONS:
Biological: Monoclonal antibody hu3S193 — Hu3S193 was to be administered intraperitoneally or intravenously at a dose of 5mg. Doses of hu3S193 were radiolabeled with 5 mCi of 111In.

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Giving monoclonal antibodies in different ways may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of monoclonal antibody therapy in treating patients who have ovarian cancer.

DETAILED DESCRIPTION:
OBJECTIVES: The primary objective iss to determine the safety of indium (111In) monoclonal antibody (mAb) hu3S193 (111In-hu3S193) given intraperitoneally or intravenously in patients with ovarian carcinoma.

Secondary objectives include comparing the localization of 111In-hu3S193 in ovarian cancer tissue after intraperitoneal vs intravenous injection and the biodistribution and pharmacokinetics of this drug when administered intraperitoneally vs intravenously in these patients as well as the formation of human anti-human antibodies (HAHA) in these patients.

OUTLINE: Patients are assigned to 1 of 2 treatment arms on a first come sequential basis. Arm I: Patients receive indium (In 111) monoclonal antibody hu3S193 (111In-hu3S193) intraperitoneally over 30 minutes. Arm II: Patients received 111In-hu3S193 intravenously (IV) over 30 minutes. Patients were to undergo surgical debulking 3-7 days following In 111In-hu3S193 administration, and biopsy samples obtained to assess radioactive uptake. Immunohistochemistry was also to be performed. Blood samples were to be obtained to assess serum radioactivity. Whole body imaging was tp be performed 3 hours after infusion of radiolabeled monoclonal antibody, on the day of surgery, and at one time point in between. Patients were followed for 30 days.

PROJECTED ACCRUAL: A total of 10 patients (5 per arm) were to be accrued for this study.

ELIGIBILITY:
Inclusion Criteria

Cytologic or pathologic diagnosis consistent with ovarian carcinoma. Scheduled to undergo surgical evaluation. Karnofsky performance status of > 60%.

Adequate organ function as defined by:

* Absolute neutrophil count (ANC) > 1.5 x 10^9/L
* Platelet count > 100 x 10^9/L
* Bilirubin < 2.0 mg/dL
* Aspartate aminotransferase (AST) and Alanine transaminase (ALT) < 2.5 X upper limit of normal
* Serum creatinine < 2.0 mg/dL
* Forced expiratory volume at one second (FEV1) and forced vital capacity (FVC)> 70% of predicted
* Left Ventricular Ejection Fraction >50%

Recovered from the toxicity of any prior therapy. No evidence of active infection which requires antibiotic therapy. > 18 years of age. Able to sign written informed consent.

Exclusion Criteria

Any significant intercurrent medical problems which may limit the amount of antibody they can tolerate, or render them ineligible for surgery.

Clinically significant cardiac disease (New York Heart Association Class III/IV, or abnormalities on ECG that are considered by the investigator to place the patient at increased risk), severe debilitating pulmonary disease, active infections or coagulation disorders.

Survival expectancy less than 12 weeks. History of autoimmune hepatitis or history of autoimmune disease. Chemotherapy, radiotherapy, or immunotherapy within four weeks prior to receiving hu3S193.

Psychiatric, addictive or other disorders that compromise the ability to give informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — ovarian carcinoma patients
Enrollment: 1 (Actual)
Dates: Start 2000-08-02 (Actual); Primary Completion 2002-02-26 (Actual); Study Completion 2002-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chaitanya R. Divgi, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intraperitoneal (IP) Infusion of 111In-hu3S193: Hu3S193 was administered intraperitoneally (IP) at a dose of 5 mg radiolabeled with 5 millicurie (mCi) of 111In.
  Patients received 10 mCi 99mTc-sulphur colloid IP administered in 500 ml of normal saline to assure the absence of any loculation or heterogeneous distribution of radioactivity in the peritoneal cavity. A paracentesis catheter was inserted and the hu3S193 was diluted in 100 mL of 5% human serum albumin and administered as a continuous intraperitoneal infusion over 30 minutes. This was followed immediately by 900 mL of normal saline.
Period: Overall Study
Arm/Group | Intraperitoneal (IP) Infusion of 111In-hu3S193 | Intravenous Infusion of 111In-hu3S193
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The 1 patient who entered the study.
Groups:
- Intraperitoneal (IP) Infusion of 111In-hu3S193: Hu3S193 was administered intraperitoneally at a dose of 5 mg radiolabeled with 5 mCi of 111In.
  Patients received 10 mCi 99mTc-sulphur colloid IP administered in 500 ml of normal saline to assure the absence of any loculation or heterogeneous distribution of radioactivity in the peritoneal cavity. A paracentesis catheter was inserted and the hu3S193 was diluted in 100 mL of 5% human serum albumin and administered as a continuous intraperitoneal infusion over 30 minutes. This was followed immediately by 900 mL of normal saline.
- Intravenous Infusion of 111In-hu3S193: Hu3S193 was to be administered intravenously at a dose of 5 mg radiolabeled with 5 mCi of 111In, diluted in 100 mL of 5% human serum albumin and administered over a 30 minute period.
- Total: Total of all reporting groups
Arm/Group | Intraperitoneal (IP) Infusion of 111In-hu3S193 | Intravenous Infusion of 111In-hu3S193 | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Grade 3 Adverse Events
Description: All toxicities were to be graded according to the Common Toxicity Criteria (CTC) Scale, version 2.0, March 1998.The study was to be terminated upon the occurrence of an adverse event of Grade 3 or greater severity that is considered definitely related to hu3S193.
Time Frame: up to 30 days
Population: The 1 patient who entered the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Intraperitoneal (IP) Infusion of 111In-hu3S193 | Intravenous Infusion of 111In-hu3S193
Number analyzed (Participants) | 1 | 0
Participants | 0 |

ADVERSE EVENTS:
Time Frame: up to 30 days
Description: All adverse events were to be recorded on the patient's case report form. All toxicities were to be graded according to the Common Toxicity Criteria (CTC) Scale, version 2.0, March 1998.
Arm/Group | Intraperitoneal (IP) Infusion of 111In-hu3S193 | Intravenous Infusion of 111In-hu3S193
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No